CLINICAL TRIAL: NCT03955354
Title: A Phase II Study of PD-1 Antibody SHR-1210 Combined With Apatinib of First-line Treatment of Advanced Acral Melanoma
Brief Title: PD-1 Antibody SHR-1210 Combined With Apatinib of First-line Treatment of Advanced Acral Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Guo, Associate Director of Peking University Cancer Hospital, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-APTN-IIT-MM
Record Dates: First submitted 2019-05-12; First posted 2019-05-20 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental arm (Experimental): SHR1210 plus apatinib
  Interventions: Drug: SHR1210; Drug: apatinib mesylate

INTERVENTIONS:
Drug: SHR1210 — SHR-1210 is a humanized anti-PD1 IgG4 monoclonal antibody
Drug: apatinib mesylate — apatinib Mesylate is a small molecule tyrosine kinase inhibitor,Through selectively inhibiting the tyrosine kinase activity of the vascular endothelial growth factor receptor 2 (VEGFR-2).

SUMMARY:
the investigators launched this exploratory study to evaluate the objective response rate (ORR) of SHR-1210 combined with apatinib mesylate in the first-line treatment of patients with advanced acral melanoma.

ELIGIBILITY:
Inclusion Criteria:

1. age:18-75 years, male or female.
2. Histopathologically confirmed recurrence, inoperable resection or metastatic acral melanoma (stage III/IV).
3. Has not received any systematic anti-tumor drug treatment.
4. Measurable disease based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
5. ECOG 0-1.
6. Adequate organ function.
7. Life expectancy of greater than 12 weeks.
8. Patient has given written informed consent.

Exclusion Criteria:

1. Patients who have or are currently undergoing additional chemotherapy, radiation therapy, targeted therapy or immunotherapy.
2. Known history of hypersensitivity to macromolecular protein preparation or any components of the SHR- 1210 formulation.
3. Subjects before or at the same time with other malignant tumors (except which has cured skin basal cell carcinoma and cervical carcinoma in situ);
4. Subjects with any active autoimmune disease or history of autoimmune disease
5. Uncontrolled clinically significant heart disease, including but not limited to the following: (1) > NYHA II congestive heart failure; (2) unstable angina, (3) myocardial infarction within the past 1 year; (4) clinically significant supraventricular arrhythmia or ventricular arrhythmia requirement for treatment or intervention;
6. Active infection or an unexplained fever > 38.5°C during screening or before the first scheduled day of dosing (subjects with tumor fever may be enrolled at the discretion of the investigator);
7. Received a live vaccine within 4 weeks of the first dose of study medication.
8. Pregnancy or breast feeding.
9. Decision of unsuitableness by principal investigator or physician-in charge.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-03-05 (Actual); Primary Completion 2020-04-10 (Estimated); Study Completion 2021-04-10 (Estimated)

PRIMARY OUTCOMES:
ORR | Time Frame: Through study completion, an average of 1 year
  Objective Response Rate

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Guo Jun, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Wang X, Wu X, Yang Y, Xu W, Tian H, Lian B, Chi Z, Si L, Sheng X, Kong Y, Zhou L, Mao L, Li S, Tang B, Yan X, Bai X, Guo J, Cui C. Apatinib combined with camrelizumab in advanced acral melanoma patients: An open-label, single-arm phase 2 trial. Eur J Cancer. 2023 Mar;182:57-65. doi: 10.1016/j.ejca.2022.12.027. Epub 2023 Jan 12. PMID 36753834
- [Derived] Tian H, Wang X, Lian B, Yan X, Si L, Chi Z, Sheng X, Kong Y, Mao L, Bai X, Tang B, Li S, Zhou L, Cui C, Guo J. Safety Profile of Immunotherapy Combined With Antiangiogenic Therapy in Patients With Melanoma: Analysis of Three Clinical Studies. Front Pharmacol. 2021 Nov 9;12:747416. doi: 10.3389/fphar.2021.747416. eCollection 2021. PMID 34858178